CLINICAL TRIAL: NCT01636427
Title: STEMI Versus NSTEMI: a Mono Versus a Multivessel Disease?
Brief Title: STEMI Versus NSTEMI: Clinical and Angiographic Differences
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Ferrara Liberato Aldo, Associate Professor of Medicine, Federico II University
Other Study IDs: 001
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Acute Coronary Syndrome
Keywords: myocardial infarction; coronary angiography; STEMI; NSTEMI
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess differences in the risk profile and in the coronary angiographic presentation between STEMI and NSTEMI. Moreover possible relationship between myocardial infarction presentation and renal function will be investigated.

DETAILED DESCRIPTION:
Assessment of risk profile. Diabetes mellitus diagnosed when fasting blood glucose (FBG) was >= 126mg/dL or if patients were taking oral hypoglycaemic drugs or were on insulin treatment. Hypertension defined as blood pressure >= 140/90 mmHg or history of antihypertensive treatment. Hypercholesterolemia,adjudicated when cholesterol levels were >= 200 mg/dL or with patients on lipid lowering treatment. Hypertriglyceridemia adjudicated on fasting triglyceride levels>= 200 mg/dL or triglyceride-lowering therapy . Obesity, defined as BMI >= 30 kg/m2.

Patients with STEMI, who had not been previously treated with thrombolysis, and those who had been undergone to an unsuccessful thrombolysis, as well as patients with NSTEMI with a TIMI score> 3 who were immediately referred to the Cat Lab and whenever possible treated with PTCA and stenting of the culprit lesion. The other patients who were referred to Cat Lab within 48 hours from the beginning of chest pain, unless their general conditions did not strongly suggest to delay the procedure after 2 more days.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in the coronary care unit (CCU) of the Department of Clinical and Experimental Medicine at the Federico 2nd University Hospital;
* Patient with indication to angiographic study even if not immediately;
* Patients referred to CCU with the diagnosis of acute myocardial infraction (AMI), type STEMI, or NSTEMI, based on pre-admission assessment of troponin I (TpI) and myocardial band creatin kinase (CK-MB;
* Diagnosis of NSTEMI/STEMI performed according to standard criteria

Exclusion criteria:

* Patients who could not undergo angiographic study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute myocardial infarction with or without ST segment elevation.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Simone, MD, Study Director — Federico 2nd University of Naples
Locations (1):
- CCU Dipartimento Assistenziale di Clinica Medica, Naples, Italy

REFERENCES:
- [Derived] Ferrara LA, Staiano L, Di Fronzo V, Ferrara F, Sforza A, Mancusi C, de Simone G. Type of myocardial infarction presentation in patients with chronic kidney disease. Nutr Metab Cardiovasc Dis. 2015 Feb;25(2):148-52. doi: 10.1016/j.numecd.2014.11.002. Epub 2014 Nov 11. PMID 25511783
- [Derived] Ferrara LA, Russo BF, Gente R, Esposito G, Rapacciuolo A, de Simone G. STEMI and NSTEMI: a mono versus a multivessel disease? Int J Cardiol. 2013 Oct 3;168(3):2905-6. doi: 10.1016/j.ijcard.2013.03.154. Epub 2013 May 3. No abstract available. PMID 23643429